CLINICAL TRIAL: NCT03917680
Title: Evaluation of New Markers (FXII and Videocapillaroscopy) in Type 3 Angioedema
Brief Title: Evaluation of New Markers in Type 3 Angioedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Olivier Michel, Head of immuno-allergology clinic, Brugmann University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-angiodema
Record Dates: First submitted 2019-04-03; First posted 2019-04-17 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Angio Edema
MeSH Terms: conditions — Angioedema | interventions — Microscopic Angioscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Type III angioedema (Experimental): White angioedema. Positive for Factor XII mutation. No C1-inhibitors anomaly. Not caused by IEC.
  Interventions: Diagnostic Test: Factor XII dosage; Genetic: p.Thr328Lys mutation detection; Diagnostic Test: Videocapillaroscopy
- Idiopathic angioedema (Experimental): White angioedema. Negative for Factor XII mutation. No C1-inhibitors anomaly. Not caused by IEC.
  Interventions: Diagnostic Test: Factor XII dosage; Genetic: p.Thr328Lys mutation detection; Diagnostic Test: Videocapillaroscopy
- Type I or II angioedema (Experimental): White angioedema. Negative for Factor XII mutation. C1-inhibitors anomaly. Not caused by IEC.
  Interventions: Diagnostic Test: Factor XII dosage; Genetic: p.Thr328Lys mutation detection; Diagnostic Test: Videocapillaroscopy
- Post IEC (conversion enzyme inhibitors) angioedema (Experimental): White angioedema. Negative for Factor XII mutation. No C1-inhibitors anomaly. Caused by IEC.
  Interventions: Diagnostic Test: Factor XII dosage; Genetic: p.Thr328Lys mutation detection; Diagnostic Test: Videocapillaroscopy
- Histaminic angioedema (Experimental): Red angioedema.Negative for Factor XII mutation. No C1-inhibitors anomaly. Not caused by IEC.
  Interventions: Diagnostic Test: Factor XII dosage; Genetic: p.Thr328Lys mutation detection; Diagnostic Test: Videocapillaroscopy
- Control (Other): Healthy individuals, no angioedema.
  Interventions: Diagnostic Test: Videocapillaroscopy

INTERVENTIONS:
Diagnostic Test: Factor XII dosage — Factor XII (FXII, Hageman factor) will be measured in plasma. It is converted to FXIIa by an activator. The FXIIa protease cleaves a chromogenic substrate and releases p-nitroaniline (pNA), which can be measured photometrically.
  Arms: Histaminic angioedema; Idiopathic angioedema; Post IEC (conversion enzyme inhibitors) angioedema; Type I or II angioedema; Type III angioedema
Genetic: p.Thr328Lys mutation detection — Sequencing of exon 9 of franking introns of FXII, for identification of the p.Thr328Lys mutation.
  Arms: Histaminic angioedema; Idiopathic angioedema; Post IEC (conversion enzyme inhibitors) angioedema; Type I or II angioedema; Type III angioedema
Diagnostic Test: Videocapillaroscopy — It is an optical method to visualize the most superficial part of the cutaneous microcirculatory network. It provides morphological information.

SUMMARY:
Angioedema is a common condition, with multiple etiologies.

Type 3 angioedema is caused by an increase in kininogenase activity responsible for an increased production of bradykinin. In some cases, it may be associated with clotting factor 12 mutations. However, other genetic abnormalities remain to be identified.

Clinically, this angioedema type 3 is similar to types 1 and 2. The patient's vital prognosis is good if the diagnosis is made and if they have access to the appropriate treatment. Otherwise a significant morbidity is associated with it, hence the importance of being able to define a diagnostic marker.

Videocapillaroscopy might be able to highlight abnormalities in the microcirculation of patients with a clinical display of angioedema.

The purpose of this study is to highlight markers allowing to make an early diagnosis of angioedema. Functional analysis of factor XII in patients with symptoms of angioedema may be an interesting marker for diagnosis.

Microcirculation abnormalities will also be evaluated by videocapillaroscopy, which may be another indicator of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Population of patients treated within the CHU Brugmann Hospital for an angioedema (and control group of healthy individuals)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Factor XII | 24 hours
  Plasma concentration of Factor XII
Presence of p.Thr328Lys mutation | 24 hours
  Genetic analysis : sequencing of the Factor VII gene. Presence/Absence of the p.Thr328Lys mutation (single nucleotide variation inducing a missense variant).
Videocapillaroscopy result | 24 hours
  It is an optical method to visualize the most superficial part of the cutaneous microcirculatory network. It provides morphological information.The result will be classified as 'normal' or 'abnormal' by the videocapillaroscopy specialist.

CONTACTS AND LOCATIONS:
Overall Officials: Oumnia Mouna, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No